CLINICAL TRIAL: NCT01342926
Title: A Phase 2, Multi-centre, Randomised, Double-masked, Placebo-controlled, Parallel-group Study to Investigate the Safety, Tolerability, Efficacy, Pharmacokinetics and Pharmacodynamics of GSK933776 in Adult Patients With Geographic Atrophy (GA) Secondary to Age-related Macular Degeneration (AMD)
Brief Title: Clinical Study to Investigate Safety and Efficacy of GSK933776 in Adult Patients With Geographic Atrophy Secondary to Age-related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114341
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Atrophy, Geographic
Keywords: age-related macular degeneration; geographic atrophy; dry AMD
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GSK933776 3 mg/kg (Experimental): 3 mg/kg administration of GSK933776 via intravenous infusion
  Interventions: Drug: GSK933776
- GSK933776 6 mg/kg (Experimental): 6 mg/kg administration of GSK933776 via intravenous infusion
  Interventions: Drug: GSK933776
- Placebo (Placebo Comparator): Placebo via intravenous infusion
  Interventions: Drug: Placebo
- GSK933776 15 mg/kg (Experimental): 15 mg/kg administration of GSK933776 via intravenous infusion
  Interventions: Drug: GSK933776

INTERVENTIONS:
Drug: GSK933776 — GSK933776
  Arms: GSK933776 15 mg/kg; GSK933776 3 mg/kg; GSK933776 6 mg/kg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of GSK933776 in the treatment of geographic atrophy secondary to age-related macular degeneration.

DETAILED DESCRIPTION:
This is a Phase 2a proof of concept study designed to evaluate the safety and efficacy of GSK933776 for the treatment of geographic atrophy secondary to age-related macular degeneration. This is a placebo-controlled parallel-group study that is double masked.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥55 years of age inclusive
* Evidence of AMD confirmed by the presence of at least 1 druse ≥125 μm diameter
* Well-demarcated GA due to AMD of total area 1.9-17 mm2 measured in the study eye
* Best-corrected visual acuity score of ≥ 35 letters (approximately 20/200 Snellen VA equivalent or better) in the study eye

Exclusion Criteria:

* Additional eye disease in the study eye that could compromise assessment of best-corrected visual acuity or imaging of the posterior pole
* History of CNV secondary to AMD in the study eye
* Any previous treatment for AMD in the study eye, approved or investigational, with the exception of dietary supplements
* Risk of cerebrovascular disease, cerebral hemorrhage or stroke
* History of systemic autoimmune disease
* Use of platelet anti-aggregants or anti-coagulants (aspirin up to 325 mg/day is allowable, or in subjects allergic or intolerable to aspirin, clopidogrel up to 75 mg/day is allowable)
* Use of chronic corticosteroids
* Uncontrolled hypertension in spite of antihypertensive medications
* Renal or hepatic insufficiency or clinically significant anemia
* More than moderate MRI white matter changes

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2011-06-01; Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (38):
- United States (37):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Arcadia, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palm Desert, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Stuart, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, New Albany, Indiana
  - GSK Investigational Site, Leawood, Kansas
  - GSK Investigational Site, Prairie Village, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Paducah, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Northfield, New Jersey
  - GSK Investigational Site, Toms River, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, West Mifflin, Pennsylvania
  - GSK Investigational Site, Ladson, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Abilene, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Silverdale, Washington
- GSK Investigational Site, Mississauga, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a parallel-group randomized study consisted of a screening visit, where 240 participants entered the observation period (minimum of 4 months), a Baseline visit at the end of observation phase, where 191 were randomized, and was followed by the treatment period (18 months), and a follow-up visit (3 months) after last dose.
Pre-assignment Details: The total duration of participation was approximately 25 months following screening.
Groups:
- Placebo: Participants received placebo (0.9 percent sodium chloride) by intravenous (IV) infusion every 28 days for 18 months.
- GSK933776 (3 mg/kg): Participants received 3 milligram (mg)/kilogram (kg) GSK933776 by IV infusion every 28 days for 18 months.
- GSK933776 (6 mg/kg): Participants received 6 mg/kg GSK933776 by IV infusion every 28 days for 18 months.
- GSK933776 (15 mg/kg): Participants received 15 mg/kg GSK933776 by IV infusion every 28 days for 18 months.
Period: Overall Study
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Started | 46 | 46 | 48 | 51
Completed | 37 | 31 | 34 | 39
Not Completed | 9 | 15 | 14 | 12
Not completed — Adverse Event | 5 | 8 | 10 | 7
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Investigator Discretion | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK933776 3 mg/kg | GSK933776 6 mg/kg | GSK933776 15 mg/kg | Total
Number analyzed (Participants) | 46 | 46 | 48 | 51 | 191
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.3 (9.55) | 77.2 (9.09) | 77.5 (8.57) | 78.6 (7.22) | 77.2 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 26 | 27 | 109
  Male | 19 | 17 | 22 | 24 | 82
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1 | 0 | 0 | 0 | 1
  White | 45 | 46 | 48 | 51 | 190

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Area of Geographic Atrophy (GA) Assessed by Color Fundus Photographs (FP) in the Study Eye
Description: Atrophic age-related macular degeneration (AMD) also called GA is characterized by thinning of the retinal pigment epithelium (RPE) and underlying choriocapillaris, as well as overlying photoreceptors in the macula. GA was evaluated by color FP at the indicated time points: screening, 6 months, 12 months and 18 months. Change from BL: (screening, month 6, 12 or 18 value minus BL value. Note screening occurs prior to BL). Only participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Efficacy Population: all participants in the Intent-to-Treat (ITT) Population who met the protocol defined inclusion criterion for area of GA assessed by color FP in the study eye in at least one visit from screening visit through BL visit, inclusive and had data of area of GA assessed by fundus autofluorescence images in the study eye for at least 75% of the visits (>=14 visits) from post-BL treatment month 2 visit to treatment month 19 visit.
Time Frame: Baseline (BL), 6 months, 12 months and 18 months
Population: Efficacy Population. Participants who developed CNV in the study eye during the treatment period are excluded from Efficacy Population per protocol.
Measure: Mean (90% Confidence Interval); unit: square millimeter (m^2)
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 34 | 30 | 35 | 40
square millimeter (m^2)
  Screening, n=34, 30, 35, 40 | -0.52 [-0.86 to -0.17] | -0.94 [-1.30 to -0.57] | -0.99 [-1.33 to -0.65] | -0.96 [-1.28 to -0.64]
  6 months, n=34, 30, 35, 39 | 0.95 [0.61 to 1.30] | 0.88 [0.51 to 1.25] | 0.73 [0.38 to 1.07] | 0.77 [0.44 to 1.09]
  12 months, n=33, 29, 34, 40 | 1.60 [1.26 to 1.95] | 1.81 [1.43 to 2.18] | 1.83 [1.49 to 2.18] | 1.89 [1.57 to 2.21]
  18 months, n=34, 30, 32, 39 | 2.60 [2.25 to 2.95] | 2.77 [2.40 to 3.14] | 2.88 [2.53 to 3.23] | 2.99 [2.67 to 3.31]
Statistical Analysis 1: Comparison: Placebo vs GSK933776 (3 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = -0.07, 90% CI 2-sided [-0.57 to 0.43] — 6 months visit
Statistical Analysis 2: Comparison: Placebo vs GSK933776 (3 mg/kg); Test type: Superiority or Other; Median Difference (Final Values) = 0.20, 90% CI 2-sided [-0.31 to 0.71] — 12 months visit
Statistical Analysis 3: Comparison: Placebo vs GSK933776 (3 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.17, 90% CI 2-sided [-0.33 to 0.68] — 18 months visit
Statistical Analysis 4: Comparison: Placebo vs GSK933776 (6 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = -0.23, 90% CI 2-sided [-0.71 to 0.26] — 6 months visit
Statistical Analysis 5: Comparison: Placebo vs GSK933776 (6 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.23, 90% CI 2-sided [-0.26 to 0.72] — 12 months visit
Statistical Analysis 6: Comparison: Placebo vs GSK933776 (6 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.28, 90% CI 2-sided [-0.21 to 0.77] — 18 months visit
Statistical Analysis 7: Comparison: Placebo vs GSK933776 (15 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = -0.18, 90% CI 2-sided [-0.66 to 0.29] — 6 months visit
Statistical Analysis 8: Comparison: Placebo vs GSK933776 (15 mg/kg); Test type: Superiority or Other; Median Difference (Final Values) = 0.28, 90% CI 2-sided [-0.19 to 0.75] — 12 months visit
Statistical Analysis 9: Comparison: Placebo vs GSK933776 (15 mg/kg); Test type: Superiority or Other; Median Difference (Final Values) = 0.39, 90% CI 2-sided [-0.08 to 0.86] — 18 months visit

2. Primary Outcome: Number of Participants With Ocular or Non-ocular Adverse Events (AEs) During the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. It includes:1. Any abnormal laboratory test results or other safety assessments including those that worsen from Baseline, and felt to be clinically significant in the medical and scientific judgment of the Investigator 2.Exacerbation (increase in frequency/intensity) of a chronic or intermittent pre-existing condition 3. New conditions detected or diagnosed after screening visit 4. Signs, symptoms, or the clinical sequelae of a suspected interaction/suspected overdose of investigational product or a concomitant medication. AEs were presented as non-ocular and ocular AEs.
Time Frame: Up to 21 months
Population: ITT Population: all participants that completed the observation period and Baseline visit, and were subsequently randomized to treatment and were administered at least one IV dose.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 46 | 46 | 48 | 51
Participants
  Non-ocular AEs | 41 | 42 | 44 | 47
  Ocular AEs | 12 | 17 | 15 | 20

3. Primary Outcome: Number of Participants With Ocular or Non-ocular Serious Adverse Events (SAEs) During the Treatment Period
Time Frame: Up to 21 months
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 46 | 46 | 48 | 51
Participants
  Non-ocular SAEs | 8 | 11 | 9 | 12
  Ocular SAEs | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance (PCI) During the Treatment Period: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital signs included SBP and DBP of Potential Clinical Importance (PCI) at the indicated time points: Baseline, month 0, month 1, month 2, month 3, month 4, month 5, month 6, month 7, month 8, month 9, month 10, month 11, month 12, month 13, month 14, month 15, month 16, month 17, month 18, early withdrawal and at follow-up visit in sitting position. 'General' is an assessment time not relative to dosing. SBP was defined as: low: <85 millimeter of mercury (mmHg) and high: >160 mmHg and DBP was defined as: low:<45 mmHg and high: >100 mmHg. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Only categories with at least one PCI value are presented.
Time Frame: Up to 21 months
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 46 | 46 | 48 | 51
Participants
  SBP Baseline General: > CCR, n=46, 46, 48, 51 | 1 | 3 | 2 | 5
  SBP Baseline General 2:> CCR, n=46, 46, 48, 50 | 1 | 2 | 2 | 4
  SBP Baseline General 3:> CCR, n=45, 46, 48, 50 | 1 | 2 | 2 | 4
  SBP Month 0, Pre-dose:> CCR, n=46, 46, 48, 51 | 2 | 1 | 1 | 1
  SBP Month 0, 0 H:> CCR, n=46, 46, 48, 51 | 1 | 1 | 2 | 3
  SBP Month 1, Pre-dose:> CCR, n=44, 44, 44, 51 | 2 | 5 | 1 | 2
  SBP Month 1, 0 H:> CCR, n=43, 44, 44, 51 | 3 | 2 | 1 | 2
  SBP Month 2, Pre-dose:> CCR, n=44, 43, 42, 49 | 1 | 2 | 3 | 2
  SBP Month 2, 0 H:> CCR, n=44, 41, 41, 49 | 1 | 4 | 1 | 3
  SBP Month 3, Pre-dose:> CCR, n=44, 37, 42, 46 | 5 | 2 | 1 | 4
  SBP Month 3, 0 H:> CCR, n=42, 35, 40, 46 | 2 | 3 | 0 | 3
  SBP Month 4, Pre-dose:> CCR, n=43, 36, 42, 46 | 1 | 4 | 0 | 3
  SBP Month 4, 0 H:> CCR, n=43, 34, 42, 46 | 1 | 2 | 1 | 3
  SBP Month 5, Pre-dose:> CCR, n=43, 36, 40, 45 | 0 | 2 | 2 | 2
  SBP Month 5, 0 H:> CCR, n=42, 36, 39, 45 | 2 | 4 | 0 | 4
  SBP Month 6, Pre-dose:> CCR, n=43, 36, 40, 45 | 0 | 3 | 1 | 3
  SBP Month 6, 0 H:> CCR, n=42, 36, 40, 45 | 2 | 1 | 3 | 3
  SBP Month 7, Pre-dose:> CCR, n=43, 35, 40, 44 | 1 | 2 | 2 | 0
  SBP Month 7, 0 H:> CCR, n=43, 33, 40, 44 | 2 | 0 | 0 | 0
  SBP Month 8, Pre-dose:> CCR, n=42, 33, 40, 44 | 2 | 2 | 1 | 1
  SBP Month 8, 0 H:> CCR, n=41, 33, 40, 44 | 1 | 3 | 0 | 1
  SBP Month 9, Pre-dose:> CCR, n=41, 33, 40, 44 | 1 | 1 | 0 | 2
  SBP Month 9, Pre-dose:< CCR, n=41, 33, 40, 44 | 1 | 0 | 0 | 0
  SBP Month 9, 0 H:> CCR, n=41, 33, 39, 44 | 0 | 1 | 0 | 1
  SBP Month 10, Pre-dose:> CCR, n=41, 32, 40, 44 | 0 | 0 | 1 | 0
  SBP Month 10, 0 H:> CCR, n=40, 32, 40, 44 | 1 | 0 | 0 | 2
  SBP Month 11, Pre-dose:> CCR, n=41, 33, 39, 42 | 2 | 2 | 3 | 2
  SBP Month 11, 0 H:> CCR, n=40, 31, 35, 41 | 1 | 0 | 1 | 1
  SBP Month 11, 0 H:< CCR, n=40, 31, 35, 41 | 1 | 0 | 0 | 0
  SBP Month 12, Pre-dose:> CCR, n=39, 30, 38, 41 | 2 | 1 | 1 | 1
  SBP Month 12, 0 H:> CCR, n=39, 30, 38, 41 | 2 | 1 | 1 | 2
  SBP Month 13, Pre-dose:> CCR, n=38, 31, 39, 39 | 0 | 1 | 1 | 2
  SBP Month 13, 0 H:> CCR, n=38, 31, 39, 38 | 1 | 0 | 0 | 1
  SBP Month 14, Pre-dose:> CCR, n=38, 31, 36, 39 | 0 | 0 | 1 | 2
  SBP Month 14, 0 H:> CCR, n=38, 31, 36, 39 | 0 | 0 | 0 | 1
  SBP Month 15, Pre-dose:> CCR, n=37, 31, 35, 39 | 0 | 0 | 1 | 3
  SBP Month 15, 0 H:> CCR, n=37, 31, 35, 39 | 1 | 0 | 0 | 0
  SBP Month 16, Pre-dose:> CCR, n=37, 31, 35, 39 | 1 | 1 | 0 | 1
  SBP Month 16, 0 H:> CCR, n=37, 31, 35, 39 | 2 | 2 | 0 | 0
  SBP Month 17, Pre-dose:> CCR, n=38, 32, 36, 40 | 2 | 2 | 1 | 0
  SBP Month 17, 0 H:> CCR, n=37, 30, 34, 48 | 1 | 2 | 0 | 1
  SBP Month 17, 0 H:< CCR, n=37, 30, 34, 48 | 0 | 1 | 0 | 0
  SBP Month 18, General:> CCR, n=36, 31, 33, 39 | 1 | 2 | 1 | 2
  SBP Early withdrawal, :> CCR, n=8, 8, 7, 4 | 0 | 1 | 1 | 1
  SBP Follow-up:> CCR, n=39, 36, 37, 43 | 1 | 0 | 0 | 1
  DBP Month 4, 0 H:< CCR, n=43, 34, 42, 46 | 1 | 0 | 0 | 0
  DBP Month 8, 0 H:> CCR, n=41, 33, 40, 44 | 1 | 0 | 0 | 0
  DBP Month 9, Pre-dose:> CCR, n=41, 33, 40, 44 | 0 | 0 | 0 | 1
  DBP Month 11, Pre-dose:> CCR, n=41, 33, 39, 42 | 0 | 0 | 1 | 0
  DBP Month 13, Pre-dose:< CCR, n=38, 31, 39, 39 | 0 | 0 | 1 | 0

5. Primary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance (PCI) During the Treatment Period: Heart Rate (HR)
Description: Vital signs included HR of CCR at the indicated time points: Baseline, Month 0, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12, Month 13, Month 14, Month 15, Month 16, Month 17, Month 18, early withdrawal and at follow-up visit in sitting position. 'General' is an assessment time not relative to dosing. HR was defined as: low:< 40 beats per minute (bpm) and high: >100 bpm. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Only categories with at least one PCI value are presented.
Time Frame: Baseline, Month 0, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12, Month 13, Month 14, Month 15, Month 16, Month 17, Month 18, early withdrawal and at follow-up visit
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 46 | 46 | 48 | 51
Participants
  HR Month 3, Pre-dose:> CCR, n=44, 37, 42, 46 | 1 | 0 | 0 | 0
  HR Month 13, Pre-dose:> CCR, n=38, 31, 39, 39 | 0 | 0 | 1 | 0

6. Primary Outcome: Number of Participants With 12-lead Electrocardiogram (ECG) of Potential Clinical Importance (PCI)
Description: 12-lead ECG was obtained after 10 minutes rest in a supine position using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT interval corrected using the Fridericia's formula (QTcF). Abnormal-clinically significant (CS) ECG measurements are presented at indicated time points: Baseline, Month 6, Month 12, Month 18, early withdrawal and at follow-up visit. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Month 6, Month 12, Month 18, early withdrawal and at follow-up visit
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 46 | 46 | 48 | 51
Participants
  ECG:CS Baseline, n=46, 46, 48, 51 | 1 | 0 | 1 | 0
  ECG:CS Month 6, n=41, 33, 37, 44 | 0 | 0 | 1 | 3
  ECG:CS Month 12, n=41, 32, 40, 40 | 0 | 1 | 1 | 0
  ECG:CS Month 18, n=38, 30, 36, 35 | 0 | 0 | 2 | 1
  ECG:CS early withdrawal, n=7, 8, 7, 3 | 0 | 1 | 2 | 0
  ECG:CS follow-up, n=39, 37, 37, 38 | 0 | 0 | 1 | 1

7. Primary Outcome: Number of Participants With Abnormal Laboratory Parameter Values of Potential Clinical Importance (PCI)
Description: The following laboratory parameters were assessed: Hematology: Platelet Count, Red Blood Cell Count, White Blood Cell (WBC) Count, Reticulocyte Count, Hemoglobin, Hematocrit, Prothrombin time-International Normalized Ratio, Activated partial thromboplastin time, Mean corpuscular volume, Mean corpuscular haemoglobin, Mean corpuscular hemoglobin concentration, Neutrophils (ANC), Lymphocytes, Monocytes, Eosinophils, and Basophils. Clinical chemistry: Blood urea nitrogen, Potassium, Aspartate aminotransferase, Total and direct bilirubin Creatinine, Chloride, Alanine aminotransferase, Uric Acid, Glucose (fasting), Total Carbon dioxide , Gamma glutamyltransferase, Albumin, Sodium, Calcium, Alkaline phosphatase, Total Protein, and HbA1c. Urine: Specific gravity, pH, glucose, protein, blood and ketones and Microscopic examination. Only those with PCIs are displayed.
Time Frame: At any point from Baseline through follow-up visit.
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 46 | 46 | 48 | 51
Participants
  Alanine Amino Transferase (less than PCI low) | 0 | 0 | 0 | 0
  Alanine Amino Transferase (Above PCI high) | 0 | 1 | 0 | 0
  Aspartate Amino Transferase (less than PCI low) | 0 | 0 | 0 | 0
  Aspartate Amino Transferase (Above PCI high) | 1 | 0 | 0 | 0
  Calcium (less than PCI low) | 0 | 0 | 0 | 1
  Calcium (Above PCI high) | 1 | 0 | 1 | 1
  CO2 content/Bicarbonate (less than PCI low) | 10 | 4 | 9 | 6
  CO2 content/B icarbonate (AbovePCI high) | 0 | 1 | 0 | 0
  Creatinine (less than PCI low) | 0 | 0 | 0 | 0
  Creatinine (Above PCI high) | 1 | 0 | 0 | 0
  Glucose (less than PCI low) | 0 | 0 | 0 | 1
  Glucose (Above PCI high) | 11 | 17 | 9 | 10
  Potassium (less than PCI low) | 0 | 0 | 0 | 0
  Potassium (Above PCI high) | 1 | 0 | 0 | 0
  Sodium (Less than PCI low) | 2 | 2 | 0 | 1
  Sodium (Above the PCI high) | 0 | 0 | 0 | 0
  Hemoglobin (less than PCI low) | 0 | 0 | 0 | 0
  Hemoglobin (Above the PCI high) | 3 | 0 | 0 | 0
  Hematocrit (less than PCI low) | 0 | 0 | 0 | 0
  Hematocrit (Above PCI high) | 5 | 2 | 2 | 3
  Lymphocytes (less than PCI low) | 2 | 2 | 1 | 1
  Lymphocytes (Above PCI high) | 0 | 0 | 0 | 0
  Total ANC (less than PCI low) | 4 | 2 | 1 | 5
  Total ANC (Above PCI high) | 0 | 0 | 0 | 0
  Platelet count (less than PCI low) | 2 | 1 | 0 | 1
  Platelet count (Above PCI high) | 0 | 0 | 0 | 0
  WBC count (less than PCI low) | 1 | 0 | 1 | 0
  WBC count (Above PCI high) | 0 | 1 | 0 | 1

8. Primary Outcome: Number of Participants With Abnormal Magnetic Resonance Imaging (MRI)
Description: Magnetic Resonance Imaging (MRI) was used as a safety assessment to monitor for amyloid related imaging abnormalities (ARIA) events in the brain. MRIs were performed at Baseline and before dose 2, before dose 3, before dose 4, before dose 6, before dose 12, before dose 18 and at follow-up. ARIA-edema/effusions (ARIA-E) and ARIA hemosiderin deposition (ARIA-H) events at any visit are reported.
Time Frame: Month 2, Month 3, Month 4, Month 6, Month 12, Month 18 and at early withdrawal
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 46 | 46 | 48 | 51
Participants
  ARIA E | 0 | 0 | 1 | 1
  ARIA H | 2 | 4 | 6 | 4

9. Secondary Outcome: Change From Baseline in Area of GA Assessed by Fundus Autofluorescence Images (hypoAF) Corresponding to GA in Study Eye
Description: Atrophic AMD also called as GA is characterized by thinning of the retinal pigment epithelium (RPE) and underlying choriocapillaris, as well as overlying photoreceptors in the macula. GA was evaluated by fundus autofluorescence images in the study eye at the indicated time points: screening, 6 months, 12 months and at 18 months. Change from Baseline: (months 6, 12,18 value minus Baseline value, respectively. Note screening occurs before baseline). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, 6 months, 12 months and 18 months
Population: Efficacy Population
Measure: Mean (90% Confidence Interval); unit: mm^2
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 34 | 30 | 35 | 40
mm^2
  Screening, n=33, 30, 34, 40 | -0.70 [-1.02 to -0.37] | -0.62 [-0.97 to -0.28] | -0.74 [-1.06 to -0.42] | -0.74 [-1.03 to -0.44]
  6 months, n=33, 30, 34, 39 | 0.81 [0.48 to 1.13] | 0.94 [0.60 to 1.29] | 0.72 [0.40 to 1.04] | 0.94 [0.64 to 1.24]
  12 months, n=32, 29, 33, 40 | 1.33 [1.00 to 1.67] | 1.74 [1.39 to 2.09] | 1.67 [1.34 to 1.99] | 1.87 [1.58 to 2.17]
  18 months, n=33, 30, 31, 39 | 2.24 [1.91 to 2.57] | 2.65 [2.31 to 3.00] | 2.41 [2.08 to 2.73] | 3.15 [2.85 to 3.45]
Statistical Analysis 1: Comparison: Placebo vs GSK933776 (3 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.14, 90% CI 2-sided [-0.34 to 0.61] — 6 months visit
Statistical Analysis 2: Comparison: Placebo vs GSK933776 (3 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.41, 90% CI 2-sided [-0.07 to 0.89] — 12 months visit
Statistical Analysis 3: Comparison: Placebo vs GSK933776 (3 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.42, 90% CI 2-sided [-0.06 to 0.89] — 18 months visit
Statistical Analysis 4: Comparison: Placebo vs GSK933776 (6 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = -0.09, 90% CI 2-sided [-0.55 to 0.37] — 6 months visit
Statistical Analysis 5: Comparison: Placebo vs GSK933776 (6 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.33, 90% CI 2-sided [-0.13 to 0.80] — 12 months visit
Statistical Analysis 6: Comparison: Placebo vs GSK933776 (6 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.17, 90% CI 2-sided [-0.30 to 0.63] — 18 months visit
Statistical Analysis 7: Comparison: Placebo vs GSK933776 (15 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.13, 90% CI 2-sided [-0.31 to 0.57] — 6 months visit
Statistical Analysis 8: Comparison: Placebo vs GSK933776 (15 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.54, 90% CI 2-sided [0.10 to 0.99] — 12 months visit
Statistical Analysis 9: Comparison: Placebo vs GSK933776 (15 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.91, 90% CI 2-sided [0.47 to 1.36] — 18 months visit

10. Secondary Outcome: Change From Baseline in Area of Total hypoAF in Study Eye
Description: Atrophic AMD also called as GA is characterized by thinning of the retinal pigment epithelium (RPE) and underlying choriocapillaris, as well as overlying photoreceptors in the macula. GA was evaluated by fundus autofluorescence at the indicated time points: screening, 6 months, 12 months and at 18 months. Change from Baseline: (Month 6, 12, 18 value minus Baseline value, respectively. Note screening occurs before baseline). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, 6 months, 12 months and 18 months
Population: Efficacy Population
Measure: Mean (90% Confidence Interval); unit: mm^2
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 34 | 30 | 35 | 40
mm^2
  Screening, n=33, 30, 34, 40 | -0.65 [-0.95 to -0.34] | -0.63 [-0.95 to 0.31] | -0.71 [-1.01 to -0.41] | -1.20 [-1.48 to -0.92]
  6 months, n=33, 30, 34, 39 | 0.91 [0.60 to 1.21] | 1.01 [0.69 to 1.33] | 0.83 [0.53 to 1.13] | 0.84 [0.56 to 1.13]
  12 months, n=32, 29, 33, 40 | 1.44 [1.13 to 1.76] | 1.90 [1.57 to 2.22] | 1.67 [1.36 to 1.97] | 1.64 [1.36 to 1.92]
  18 months, n=33, 30, 31, 39 | 2.35 [2.04 to 2.65] | 2.67 [2.35 to 2.99] | 2.46 [2.15 to 2.77] | 2.85 [2.57 to 3.13]
Statistical Analysis 1: Comparison: Placebo vs GSK933776 (3 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.10, 90% CI 2-sided [-0.34 to 0.55] — 6 months visit
Statistical Analysis 2: Comparison: Placebo vs GSK933776 (3 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.45, 90% CI 2-sided [0.00 to 0.90] — 12 months visit
Statistical Analysis 3: Comparison: Placebo vs GSK933776 (3 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.33, 90% CI 2-sided [-0.12 to 0.77] — 18 months visit
Statistical Analysis 4: Comparison: Placebo vs GSK933776 (6 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = -0.08, 90% CI 2-sided [-0.51 to 0.35] — 6 months visit
Statistical Analysis 5: Comparison: Placebo vs GSK933776 (6 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.23, 90% CI 2-sided [-0.21 to 0.66] — 12 months visit
Statistical Analysis 6: Comparison: Placebo vs GSK933776 (6 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.12, 90% CI 2-sided [-0.32 to 0.55] — 18 months visit
Statistical Analysis 7: Comparison: Placebo vs GSK933776 (15 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = -0.06, 90% CI 2-sided [-0.48 to 0.35] — 6 months visit
Statistical Analysis 8: Comparison: Placebo vs GSK933776 (15 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.20, 90% CI 2-sided [-0.22 to 0.62] — 12 months visit
Statistical Analysis 9: Comparison: Placebo vs GSK933776 (15 mg/kg); Test type: Superiority or Other; Mean Difference (Final Values) = 0.50, 90% CI 2-sided [0.08 to 0.92] — 18 months visit

11. Secondary Outcome: Number of Participants Losing Letters in Early Treatment Diabetic Retinopathy Study (ETDRS)-Best Corrected Visual Acuity (BCVA) Score at Month 12 and Month 18 for Each Eye
Description: Participants enrolled into the study were required to have a best-corrected ETDRS visual acuity score of at least 35 letters as determined by ETDRS-BCVA evaluation. ETDRS-BCVA score was assessed at the indiated time points at: Month 12 and Month 18 with categorical changes in the number of participants losing >30, >=15, >=10, >=5 and <5 letters.
Time Frame: Month 12 and Month 18
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 46 | 46 | 48 | 51
Participants
  M12:Study eye, Losing > 30 letters | 1 | 0 | 1 | 1
  M12:Study eye, Losing >= 15 letters | 3 | 0 | 2 | 6
  M12:Study eye, Losing >= 10 letters | 4 | 1 | 3 | 9
  M12:Study eye, Losing >= 5 letters | 11 | 7 | 10 | 14
  M12:Study eye, Losing <5 | 28 | 23 | 28 | 27
  M12:fellow eye, Losing > 30 letters | 1 | 0 | 0 | 1
  M12:fellow eye, Losing >= 15 letters | 5 | 0 | 0 | 2
  M12:fellow eye, Losing >= 10 letters | 7 | 3 | 0 | 3
  M12:fellow eye, Losing >= 5 letters | 8 | 6 | 6 | 11
  M12:fellow eye, Losing <5 | 31 | 24 | 31 | 30
  M18:Study eye, Losing > 30 letters | 1 | 1 | 2 | 1
  M18:Study eye, Losing >= 15 letters | 3 | 1 | 6 | 5
  M18:Study eye, Losing >= 10 letters | 10 | 4 | 9 | 10
  M18:Study eye, Losing >= 5 letters | 15 | 10 | 11 | 12
  M18:Study eye, Losing <5 | 22 | 21 | 22 | 27
  M18:fellow eye, Losing > 30 letters | 2 | 0 | 0 | 0
  M18:fellow eye, Losing >= 15 letters | 4 | 2 | 1 | 2
  M18:fellow eye, Losing >= 10 letters | 6 | 4 | 1 | 3
  M18:fellow eye, Losing >= 5 letters | 10 | 7 | 4 | 9
  M18:fellow eye, Losing <5 | 27 | 24 | 28 | 30

12. Secondary Outcome: Mean Change in ETDRS-BCVA Score From Baseline at Every Month up to Month 18
Description: Participants enrolled into the study were required to have a best-corrected ETDRS visual acuity score of at least 35 letters as determined by ETDRS-BCVA evaluation. ETDRS-BCVA score was assessed as change from baseline in the mean best-corrected ETDRS visual acuity score at 18 months. Change from Baseline is defined as post-dose visit value minus Baseline value. Note that screening occurs before baseline. Values were truncated to one decimal place and negative sign retained where value is negative and the truncated value is zero. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and every month up to Month 18
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 46 | 46 | 48 | 51
Scores on a scale
  Study eye, screening, n=46,46,48,48 | 0.2 (5.76) | 2.6 (6.31) | 0.6 (7.69) | 0.1 (8.09)
  Study eye, month 1, n=44,44,44,44 | 0.7 (4.77) | 0.3 (5.13) | 0.4 (5.02) | -1.3 (5.14)
  Study eye, month 2, n=44,43,43,43 | -0.3 (7.09) | 1.0 (4.68) | 1.2 (4.45) | -0.3 (6.38)
  Study eye, month 3, n=43,37,42,42 | 0.0 (6.57) | 0.5 (7.53) | 1.0 (5.86) | -0.0 (6.39)
  Study eye, month 4, n=43,36,42,42 | 0.9 (7.93) | 1.6 (6.72) | 0.3 (6.00) | -1.4 (8.09)
  Study eye, month 5, n=43,36,39, 39 | -1.2 (9.03) | 0.5 (6.60) | 2.2 (4.88) | -2.6 (9.36)
  Study eye, month 6, n=43,36,40,40 | -0.8 (9.90) | 1.1 (6.91) | 1.6 (6.55) | -1.0 (7.80)
  Study eye, month 7, n=43,36,40,40 | 0.3 (10.49) | 1.4 (7.04) | 1.1 (8.35) | -1.7 (7.71)
  Study eye, month 8, n=42,33,40,40 | -0.0 (11.07) | 1.5 (5.94) | 0.6 (8.26) | -3.4 (8.87)
  Study eye, month 9, n=41,33,40,40 | -0.8 (10.90) | 1.0 (5.97) | 1.3 (7.39) | -2.2 (8.93)
  Study eye, month 10, n=41,32,40,40 | 0.0 (11.12) | -0.6 (7.40) | 0.7 (10.05) | -3.3 (9.86)
  Study eye, month 11, n=41,33,40,40 | 0.4 (11.69) | 0.1 (6.77) | -0.6 (8.87) | -4.1 (8.92)
  Study eye, month 12, n=39,30,38,38 | -1.3 (11.57) | -0.4 (6.12) | 0.3 (9.94) | -4.4 (9.69)
  Study eye, month 13, n=38,31,39,39 | 0.7 (8.21) | -0.1 (6.89) | -0.9 (9.93) | -4.2 (9.79)
  Study eye, month 14, n=38,31,35,35 | -1.3 (10.84) | -0.2 (8.12) | -1.2 (10.46) | -3.8 (9.68)
  Study eye, month 15, n=37,31,35,35 | -1.7 (11.13) | -1.7 (9.09) | -2.4 (11.33) | -4.0 (9.36)
  Study eye, month 16, n=37,31,35,35 | -0.6 (10.06) | -2.1 (8.71) | -2.2 (12.48) | -3.9 (9.83)
  Study eye, month 17, n=38,32,36,36 | -3.9 (14.56) | -1.9 (8.33) | -1.3 (11.85) | -3.9 (9.48)
  Study eye, month 18, n=37,31,33,33 | -3.0 (11.58) | -2.2 (10.61) | -3.6 (15.05) | -4.4 (9.72)
  Fellow eye, screening, n=46,45,46,51 | -0.0 (6.74) | 1.0 (8.30) | 0.7 (6.81) | 0.4 (9.46)
  Fellow eye, month 1, n=44,44,43,51 | 0.8 (5.01) | 1.6 (6.22) | 0.3 (5.52) | -0.8 (7.52)
  Fellow eye, month 2, n=44,43,42,49 | 1.1 (5.61) | 2.3 (7.21) | 1.4 (5.50) | 1.0 (8.86)
  Fellow eye, month 3, n=43,37,41,46 | 1.8 (7.73) | 2.3 (8.01) | 1.2 (6.63) | 2.0 (6.57)
  Fellow eye, month 4, n=43,36,41,46 | 2.7 (8.32) | 3.6 (7.80) | 2.6 (7.95) | 1.1 (6.63)
  Fellow eye, month 5, n=43,36,38,46 | 2.4 (8.13) | 3.6 (9.47) | 1.5 (8.01) | 1.8 (5.79)
  Fellow eye, month 6, n=43,36,39,43 | 0.4 (11.62) | 3.2 (8.81) | 3.4 (6.55) | 2.8 (7.66)
  Fellow eye, month 7, n=43,36,39,44 | 0.4 (13.15) | 3.5 (8.70) | 3.3 (7.01) | 1.9 (6.24)
  Fellow eye, month 8, n=42,33,39,44 | -0.4 (14.53) | 3.2 (7.08) | 1.2 (7.75) | 2.6 (8.16)
  Fellow eye, month 9, n=41,33,39,44 | -0.8 (12.42) | 4.5 (7.12) | 2.7 (7.28) | 3.0 (7.59)
  Fellow eye, month 10, n=41, 32,39,44 | -0.8 (14.22) | 4.2 (7.58) | 2.4 (8.61) | 1.2 (9.26)
  Fellow eye, month 11, n=41,33,39,42 | 0.1 (12.57) | 2.5 (7.96) | 1.0 (9.05) | 2.7 (7.89)
  Fellow eye, month 12, n=39,30,37,41 | -0.9 (13.48) | 3.2 (8.58) | 2.7 (7.36) | 0.5 (10.34)
  Fellow eye, month 13, n=38,31,37,39 | -0.2 (13.62) | 3.7 (7.92) | 1.8 (7.15) | 2.1 (8.64)
  Fellow eye, month 14, n=38,31,34,39 | -0.3 (13.22) | 1.8 (11.85) | 2.9 (7.65) | 1.9 (7.69)
  Fellow eye, month 15, n=37,31,34,39 | -1.2 (13.44) | 1.7 (8.13) | 2.3 (7.28) | 2.3 (6.45)
  Fellow eye, month 16, n=37,31,34,39 | 0.1 (12.27) | 2.0 (9.42) | 2.9 (8.42) | 2.4 (7.88)
  Fellow eye, month 17, n=38,32,35,40 | -2.1 (13.53) | 2.7 (9.55) | 1.6 (9.32) | 1.6 (8.58)
  Fellow eye, month 18, n=37,31,32,39 | -1.1 (13.12) | 1.2 (10.01) | 2.5 (8.98) | 0.4 (8.04)

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the End of Dosing Interval at Steady-state (AUC0-28d) of GSK933776 in Geographic Atrophy Participants
Description: Area under the plasma concentration-time curve from time 0 to the end of dosing interval at steady-state; derived from dose and clearance parameters was evaluated. Blood samples were collected at the indicated time points on Day 56, Day 63, 70 or 77, Day 84, Day 112, Day 140, Day 224, Day 308, Day 392 and Day 476.
Time Frame: Day 56, Day 63, 70 or 77, Day 84, Day 112, Day 140, Day 224, Day 308, Day 392 and Day 476
Population: Pharmacokinetic (PK) Parameter Population: all participants in the ITT Population with derived PK parameters
Measure: Geometric Mean (95% Confidence Interval); unit: microgram (mcg)*hours (h)/mL
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 0 | 42 | 43 | 49
microgram (mcg)*hours (h)/mL |  | 16725.96 [15814.25 to 17690.24] | 29717.17 [28241.55 to 31269.90] | 69485.24 [66687.22 to 72400.66]

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) and Pre-dose (Trough) Concentration at the End of the Dosing Interval (Ctau) of GSK933776 in Geographic Atrophy Participants
Description: Blood samples were collected at the indicated time points on Day 56, Day 63, 70 or 77, Day 84, Day 112, Day 140, Day 224, Day 308, Day 392 and Day 476
Time Frame: Day 56, Day 63, 70 or 77, Day 84, Day 112, Day 140, Day 224, Day 308, Day 392 and Day 476
Population: PK Parameter Population
Measure: Geometric Mean (95% Confidence Interval); unit: nanogram (ng)/mL
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 0 | 42 | 43 | 49
nanogram (ng)/mL
  Cmax |  | 82311.15 [73272.43 to 92464.87] | 142728.2 [126308.3 to 161282.8] | 350716.9 [314882.9 to 390628.9]
  Ctau |  | 8551.70 [7565.08 to 9667.00] | 15512.19 [13721.27 to 17536.86] | 37589.25 [33641.86 to 41999.82]

15. Secondary Outcome: Clearance (CL) of GSK933776 in Geographic Atrophy Participants
Description: as for outcome 14
Time Frame: Day 56, Day 63, 70 or 77, Day 84, Day 112, Day 140, Day 224, Day 308, Day 392 and Day 476
Population: PK Parameter Population
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 0 | 42 | 43 | 49
mL/h |  | 14.66 [13.87 to 15.49] | 14.90 [13.93 to 15.94] | 16.09 [15.16 to 17.08]

16. Secondary Outcome: Estimation of Terminal Phase Half-life (T1/2) of GSK933776 in Geographic Atrophy Participants
Description: as for outcome 14
Time Frame: Day 56, Day 63, 70 or 77, Day 84, Day 112, Day 140, Day 224, Day 308, Day 392 and Day 476
Population: PK Parameter Population
Measure: Geometric Mean (95% Confidence Interval); unit: Days
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 0 | 42 | 43 | 49
Days |  | 11.67 [11.37 to 11.98] | 11.87 [11.52 to 12.24] | 11.27 [10.93 to 11.62]

17. Secondary Outcome: Volume of Distribution at Steady-state (Vdss) of GSK933776 in Geographic Atrophy Participants Estimated From Population PK Modeling
Description: as for outcome 14
Time Frame: Day 56, Day 63, 70 or 77, Day 84, Day 112, Day 140, Day 224, Day 308, Day 392 and Day 476
Population: PK Parameter Population
Measure: Geometric Mean (95% Confidence Interval); unit: mL
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 0 | 42 | 43 | 49
mL |  | 5618.72 [5417.37 to 5827.55] | 5825.03 [5569.75 to 6092.02] | 5959.42 [5730.63 to 6197.35]

18. Secondary Outcome: The Pharmacodynamic Effects of GSK933776 Total (Bound and Unbound) Plasma Total Amyloid Beta (Abeta42), and Amyloid Beta Fragments (Abeta18-35), if Possible, Unbound Plasma Aβ Fragments (Abeta1-22)
Description: Blood samples were collected at the indicated time points on Baseline, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15 and Month 18. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15 and Month 18
Population: PD Concentration Population: all participants in the ITT Population with at least one PD sample
Measure: Mean (Standard Deviation); unit: picogram (PG)/ML
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Number analyzed (Participants) | 46 | 44 | 48 | 51
picogram (PG)/ML
  Ab1-22 Baseline, n=45,42,46,48 | 715.69 (237.06) | 702.63 (278.771) | 729.12 (260.094) | 709.04 (205.697)
  Ab1-22 month 3, PD, n=41,39,39, 46 | 675.95 (158.88) | 833.22 (557.283) | 721.04 (436.777) | 756.85 (367.050)
  Ab1-22, month 3, 1H post, n=40,39,36,44 | 706.74 (159.38) | 101.59 (88.045) | 86.57 (76.641) | 73.29 (115.732)
  Ab1-22, month 3, 3H post, n=40,39,37,43 | 707.00 (168.67) | 142.63 (144.798) | 92.22 (80.565) | 67.42 (50.512)
  Ab1-22, month 3, 7 D post M3, n=9,12,14,9 | 701.59 (232.76) | 571.23 (445.822) | 438.53 (270.154) | 274.57 (190.397)
  Ab1-22, month 3, 14 D post M3, n=9,9,6,14 | 825.32 (197.52) | 587.33 (364.383) | 357.47 (228.729) | 444.97 (149.504)
  Ab1-22, month 3, 21 D post M3, n=23,15, 18,22 | 592.13 (205.75) | 669.63 (377.229) | 730.61 (419.034) | 674.38 (270.355)
  Ab1-22 month 4, PD, n=39,32,39,44 | 671.16 (207.78) | 798.93 (588.940) | 763.67 (468.654) | 811.97 (300.797)
  Ab1-22, month 4, 1 H post, n=38,30,37,42 | 681.64 (245.28) | 95.12 (101.607) | 114.68 (142.473) | 57.27 (33.590)
  Ab1-22, month 4, 3 H post, n=38,31,35,41 | 713.41 (213.60) | 113.68 (120.182) | 104.79 (85.438) | 64.05 (36.625)
  Ab1-22 month 5, PD, n=38,29,38,46 | 686.71 (242.20) | 876.62 (587.141) | 725.24 (432.365) | 829.03 (374.933)
  Ab1-22, month 5, 1 H post, n=38,30,37,43 | 671.58 (263.41) | 106.23 (117.776) | 113.36 (114.519) | 52.91 (31.684)
  Ab1-22, month 5, 3 H post, n=38,29,36,43 | 680.31 (233.46) | 131.86 (128.104) | 99.54 (87.204) | 93.08 (227.209)
  Ab1-22 month 6, PD, n=36,31,35,45 | 664.05 (286.35) | 944.83 (666.482) | 786.00 (395.099) | 796.74 (321.794)
  Ab1-22, month 6, 1 H post, n=35,30,32,43 | 745.27 (262.59) | 98.90 (89.639) | 87.87 (76.150) | 60.33 (45.976)
  Ab1-22, month 6, 3 H post, n=36,30,31,43 | 717.93 (255.49) | 127.41 (114.486) | 101.20 (79.938) | 93.26 (209.024)
  Ab1-22 month 9, PD, n=38,28,34,42 | 698.54 (231.31) | 965.46 (664.425) | 731.34 (460.298) | 710.63 (313.891)
  Ab1-22, month 9, 1 H post, n=37,28,34,41 | 749.19 (230.82) | 187.83 (206.605) | 93.58 (103.359) | 51.96 (33.876)
  Ab1-22, month 9, 3 H post, n=37,26,34,40 | 706.89 (259.60) | 172.30 (159.749) | 101.28 (103.129) | 54.65 (36.712)
  Ab1-22 month 12, PD, n=38,30,37,41 | 688.50 (183.35) | 980.25 (342.607) | 724.92 (366.266) | 669.94 (417.194)
  Ab1-22, month 12, 1 H post, n=37,30,34,38 | 687.88 (203.57) | 87.34 (74.521) | 68.86 (77.852) | 55.36 (46.136)
  Ab1-22, month 12, 3 H post, n=37,31,31,37 | 680.21 (221.73) | 162.41 (231.741) | 79.92 (78.323) | 56.04 (48.351)
  Ab1-22 month 15, PD, n=36,27,31,39 | 667.13 (279.48) | 1011.37 (458.087) | 877.55 (589.463) | 451.65 (310.992)
  Ab1-22, month 15, 1 H post, n=38,28,32,38 | 674.94 (272.43) | 102.84 (69.049) | 92.10 (109.355) | 52.10 (89.673)
  Ab1-22, month 15, 3 H post, n=36,27,29,36 | 664.14 (321.47) | 135.58 (78.565) | 120.82 (124.908) | 54.85 (76.984)
  Ab1-22 month 18, PD, n=35,28,34,38 | 562.41 (186.57) | 1019.37 (510.656) | 968.23 (582.016) | 396.39 (324.875)
  Ab1-22, month 18, 1 H post, n=35,27,33,37 | 603.70 (184.05) | 94.79 (54.323) | 93.83 (77.725) | 42.40 (37.672)
  Ab1-22, month 18, 3 H post, n=34,26,32,37 | 572.09 (161.77) | 127.62 (67.299) | 103.38 (84.009) | 38.60 (22.256)
  Ab 18-34 Baseline, n=43,37,45,38 | 743.82 (380.653) | 819.49 (296.673) | 743.81 (406.171) | 579.25 (277.483)
  Ab 18-34 month 3, PD, n=39,38,37,45 | 785.65 (454.869) | 18592.94 (5597.893) | 27957.34 (8921.484) | 33131.16 (11098.580)
  Ab 18-34, month 3, 1H post, n=39,38,33,43 | 1408.61 (3774.763) | 22652.19 (6213.219) | 31669.84 (9225.846) | 34207.81 (11060.95)
  Ab 18-34, month 3, 3H post, n=37,38,32,43 | 836.20 (429.027) | 26215.58 (7838.227) | 34779.13 (9115.431) | 38141.47 (9668.57)
  Ab 18-34, month 3, 7 D post M3, n=7,11,11,8 | 922.92 (370.492) | 44763.87 (6895.501) | 56154.01 (13944.00) | 49791.95 (16363.48)
  Ab 18-34, month 3, 14 D post M3, n=9,11,4,14 | 1068.33 (779.813) | 35763.55 (6062.090) | 38729.93 (7646.892) | 41809.21 (12065.52)
  Ab 18-34, month 3, 21 D post M3, n=18,15,16,20 | 811.92 (321.961) | 21020.41 (9021.023) | 35400.30 (7979.633) | 43914.27 (11231.62)
  Ab 18-34 month 4, PD, n=35,31,35, | 894.86 (443.914) | 17268.05 (5857.907) | 26716.77 (10948.73) | 33334.70 (8458.286)
  Ab 18-34, month 4, 1 H post, n=32,31,33,41 | 885.66 (377.125) | 20994.88 (6978.372) | 29940.66 (10073.83) | 34964.84 (10002.35)
  Ab 18-34, month 4, 3 H post, n=32,31,31,40 | 881.00 (347.112) | 24894.01 (7706.804) | 32626.1 (10801.42) | 37516.27 (10955.53)
  Ab 18-34 month 5, PD, n=33,28,35, 46 | 951.92 (516.887) | 18728.68 (6760.913) | 27358.59 (11742.90) | 32652.34 (9462.231)
  Ab 18-34, month 5, 1 H post, n=34,28,35,42 | 962.84 (490.933) | 23681.97 (7190.390) | 29660.64 (10276.52) | 33182.12 (9115.903)
  Ab 18-34, month 5, 3 H post, n=36,28,34,40 | 893.16 (485.544) | 25711.80 (6767.509) | 33735.73 (12433.44) | 34169.47 (8984.387)
  Ab 18-34 month 6, PD, n=34,29,35,45 | 838.42 (425.702) | 18801.95 (7605.319) | 30073.49 (11286.35) | 32538.92 (8469.383)
  Ab 18-34, month 6, 1 H post, n=33,28,33,43 | 1566.28 (4065.365) | 22511.14 (7848.044) | 33259.36 (10975.41) | 34146.93 (10421.73)
  Ab 18-34, month 6, 3 H post, n=32,29,32,42 | 846.19 (421.980) | 26457.65 (7860.423) | 37724.75 (12990.61) | 37139.56 (12656.18)
  Ab 18-34 month 9, PD, n=33,22,33,42 | 609.41 (329.151) | 18187.69 (6942.978) | 27101.57 (11334.69) | 33653.88 (12115.89)
  Ab 18-34, month 9, 1 H post, n=33,23,32,40 | 617.63 (339.050) | 22315.06 (8256.360) | 29347.65 (11567.85) | 34807.59 (11458.57)
  Ab 18-34, month 9, 3 H post, n= | 1503.09 (4809.095) | 26238.37 (8950.567) | 31788.45 (12230.14) | 37923.17 (13928.32)
  Ab 18-34 month 12, PD, n=32,22,33,39 | 565.11 (269.418) | 15213.11 (7350.114) | 24193.39 (10117.95) | 33105.49 (9358.291)
  Ab 18-34, month 12, 1 H post, n=37,29,36,40 | 555.39 (296.989) | 21439.13 (9174.242) | 25724.20 (9073.725) | 35273.76 (11497.23)
  Ab 18-34, month 12, 3 H post, n=35,29,33,37 | 1532.25 (5463.999) | 21295.72 (6471.001) | 28771.21 (9392.402) | 37831.60 (11953.37)
  Unscheduled, n=0,0,0,1 | NA (NA) — NA indicates that no data is available for those Arms - only one sample for one participant was collected at the 'Unscheduled' time point. | NA (NA) — NA indicates that no data is available for those Arms - only one sample for one participant was collected at the 'Unscheduled' time point. | NA (NA) — NA indicates that no data is available for those Arms - only one sample for one participant was collected at the 'Unscheduled' time point. | 18312.40 (NA) — NA indicates that the SD is not available due to only 1 participant analyzed.
  Ab 18-34 month 15, PD, n=35,26,30,37 | 461.47 (414.780) | 16852.93 (6707.423) | 22121.87 (7510.438) | 28887.86 (7891.499)
  Ab 18-34, month 15, 1 H post, n=30,27,31,37 | 530.88 (392.825) | 20158.76 (7147.691) | 26219.44 (7873.201) | 28914.08 (9757.638)
  Ab 18-34, month 15, 3 H post, n=26,25,30,33 | 825.72 (1527.743) | 23509.29 (9303.296) | 29785.49 (9191.623) | 31653.02 (8909.182)
  Ab 18-34 month 18, PD, n=27,27,34,38 | 3144.40 (9209.436) | 14266.65 (7931.78) | 21134.85 (8638.106) | 28107.98 (9780.376)
  Ab 18-34, month 18, 1 H post, n=28,27,33,37 | 2988.76 (8357.739) | 18503.81 (9250.829) | 24124.61 (7723.055) | 29913.96 (10878.95)
  Ab 18-34, month 18, 3 H post, n=28,27,32,36 | 3144.44 (9129.569) | 21691.51 (8999.993) | 28580.63 (8684.780) | 31441.25 (10084.47)
  Ab42 Baseline, n=38,39,41,20 | 139.90 (173.673) | 92.27 (79.938) | 99.86 (85.958) | 384.28 (760.175)
  Ab42 month 3, PD, n=36,38,40, 37 | 167.67 (255.009) | 988.18 (370.001) | 1523.72 (662.292) | 1689.03 (652.829)
  Ab42, month 3, 1H post, n= 35,38,37,37 | 145.58 (230.115) | 1152.92 (420.811) | 1589.49 (629.616) | 1778.93 (644.677)
  Ab42, month 3, 3H post, n=36,38,38,35 | 207.98 (345.712) | 1296.12 (438.252) | 1672.97 (664.08) | 1959.40 (707.293)
  Ab42, month 3, 7 D post M3, n=9,11,15,6 | 77.61 (34.043) | 1697.51 (401.839) | 2022.63 (897.848) | 2007.92 (673.666)
  Ab42, month 3, 14 D post M3, n=8,11,6,9 | 244.51 (277.941) | 1599.87 (373.006) | 1608.36 (360.506) | 1695.08 (234.094)
  Ab42, month 3, 21 D post M3, n=18,14, 18,19 | 169.91 (368.921) | 1015.81 (394.872) | 1559.20 (469.99) | 2096.98 (769.107)
  Ab42 month 4, PD, n=35,33,39, 29 | 195.41 (331.409) | 984.70 (329.701) | 1381.96 (666.242) | 1575.82 (606.059)
  Ab42, month 4, 1 H post, n=33,33,36,30 | 202.80 (338.066) | 1095.62 (348.452) | 1541.21 (657.964) | 1821.73 (817.436)
  Ab42, month 4, 3 H post, n=35,32,33,30 | 201.34 (334.588) | 1313.46 (457.509) | 1714.54 (689.400) | 1744.84 (768.485)
  Ab42 month 5, PD, n=33,32,39,34 | 186.73 (316.028) | 978.6 (403.364) | 1422.10 (620.253) | 1450.71 (599.032)
  Ab42, month 5, 1 H post, n=33,32,40,32 | 182.94 (293.746) | 1214.53 (409.266) | 1526.11 (651.944) | 1572.92 (565.403)
  Ab42, month 5, 3 H post, n=32,31,39,31 | 177.67 (285.526) | 1351.07 (416.735) | 1755.13 (741.876) | 1696.91 (708.505)
  Ab42 month 6, PD, n=27,30,38,33 | 218.22 (418.144) | 1074.00 (495.245) | 1711.71 (1502.526) | 1509.95 (425.854)
  Ab42, month 6, 1 H post, n=29,30,36,32 | 233.29 (401.633) | 1241.12 (528.261) | 1835.47 (1447.740) | 1613.65 (493.896)
  Ab42, month 6, 3 H post, n=27,32,34,31 | 222.86 (435.218) | 1421.14 (545.844) | 2074.12 (1509.886) | 1723.03 (790.928)
  Ab42 month 9, PD, n=19,27,37,38 | 191.73 (243.600) | 1049.44 (419.011) | 1650.02 (1809.009) | 1519.98 (842.690)
  Ab42, month 9, 1 H post, n=18,27,35,38 | 179.70 (212.048) | 1218.78 (390.582) | 1723.09 (1521.428) | 1591.82 (749.909)
  Ab42, month 9, 3 H post, n=17,24,36,37 | 201.73 (238.311) | 1420.29 (486.511) | 1857.20 (1642.287) | 1691.34 (854.596)
  Ab42 month 12, PD, n=13,27,37,37 | 200.69 (265.476) | 916.06 (451.841) | 1253.07 (566.682) | 1221.73 (504.928)
  Ab42, month 12, 1 H post, n=14,26,33,34 | 190.76 (246.820) | 1211.53 (488.773) | 1383.67 (605.187) | 1324.37 (598.120)
  Ab42, month 12, 3 H post, n=15,27,30,34 | 193.7 (240.465) | 1238.51 (478.369) | 1489.97 (519.535) | 1411.51 (593.534)
  Ab42 month 15, PD, n=11,27,30,37 | 255.38 (510.410) | 1022.33 (415.974) | 1109.96 (467.439) | 1157.26 (347.208)
  Ab42, month 15, 1 H post, n=11,27,34,36 | 241.82 (469.544) | 1181.69 (458.696) | 1266.70 (430.670) | 1172.10 (300.788)
  Ab42, month 15, 3 H post, n=10,26,30,34 | 272.83 (524.796) | 1360.57 (510.374) | 1488.49 (479.831) | 1257.99 (330.407)
  Ab42 month 18, PD, n=8,29,29,36 | 127.77 (106.936) | 722.52 (381.288) | 997.11 (438.328) | 1087.18 (270.541)
  Ab42, month 18, 1 H post, n=10,28,29,35 | 119.29 (95.689) | 900.42 (434.525) | 1134.77 (439.660) | 1205.27 (389.468)
  Ab42, month 18, 3 H post, n=10,28,27,35 | 109.09 (88.111) | 1024.30 (472.320) | 1326.97 (491.829) | 1254.63 (304.826)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication up to approximately 21 months.
Description: SAEs and non-serious AEs were collected in members of the ITT Population, comprised of participants that completed the observation period and Baseline visit, and were subsequently randomized to treatment and were administered at least one IV dose.
Arm/Group | Placebo | GSK933776 (3 mg/kg) | GSK933776 (6 mg/kg) | GSK933776 (15 mg/kg)
Serious Adverse Events (participants affected / at risk) | 9/46 | 11/46 | 9/48 | 12/51
Other Adverse Events (participants affected / at risk) | 31/46 | 37/46 | 32/48 | 37/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | GSK933776 (3 mg/kg) (N=46) | GSK933776 (6 mg/kg) (N=48) | GSK933776 (15 mg/kg) (N=51)
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary ostial stenosis (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Subendocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular asystole (Cardiac disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Orthostatic hypertension (Vascular disorders) | 0 | 1 | 0 | 0
vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | GSK933776 (3 mg/kg) (N=46) | GSK933776 (6 mg/kg) (N=48) | GSK933776 (15 mg/kg) (N=51)
Urinary tract infection (Infections and infestations) | 3 | 6 | 4 | 1
Bronchitis (Infections and infestations) | 5 | 2 | 2 | 3
Sinusitis (Infections and infestations) | 6 | 1 | 1 | 3
Nasopharyngitis (Infections and infestations) | 3 | 3 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 0 | 1
Retinal haemorrhage (Eye disorders) | 3 | 4 | 3 | 4
Blepharitis (Eye disorders) | 2 | 5 | 4 | 1
Visual acuity reduced (Eye disorders) | 2 | 3 | 1 | 1
Vitreous detachment (Eye disorders) | 1 | 3 | 1 | 1
Macular fibrosis (Eye disorders) | 0 | 0 | 1 | 3
Headache (Nervous system disorders) | 1 | 4 | 4 | 3
Dizziness (Nervous system disorders) | 2 | 3 | 3 | 2
Nerve compression (Nervous system disorders) | 0 | 3 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 3 | 0 | 0
Oedema peripheral (General disorders) | 2 | 3 | 1 | 4
Peripheral swelling (General disorders) | 3 | 1 | 0 | 2
Fatigue (General disorders) | 0 | 3 | 2 | 0
Oedema (General disorders) | 0 | 3 | 1 | 0
Pyrexia (General disorders) | 0 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3
Nausea (Gastrointestinal disorders) | 2 | 4 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1 | 4
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 4
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 4
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 3
Ventricular extrasystoles (Cardiac disorders) | 0 | 2 | 2 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 3 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 1 | 3
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 1
Depression (Psychiatric disorders) | 4 | 0 | 2 | 2
Insomnia (Psychiatric disorders) | 3 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 2 | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1
Cardiac murmur (Investigations) | 1 | 4 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 2 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.